CLINICAL TRIAL: NCT05769023
Title: A Spatial Analysis of Hotspots and Targeted Injection Settings Pilot Intervention for HIV Prevention Among People Who Inject Drugs in Baltimore, Maryland, Supplement
Brief Title: A Spatial Analysis of Hotspots and Targeted Injection Settings Pilot Intervention for HIV Prevention Among People Who Inject Drugs
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 5R01DA050470S1; IRB00019139 (Other: JHSPH IRB); 5R01DA050470 (NIH)
Record Dates: First submitted 2023-03-01; First posted 2023-03-15 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: pilot of an intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): behavioral intervention
  Interventions: Behavioral: Intervention test

INTERVENTIONS:
Behavioral: Intervention test — behavioral sessions to promote vaccines

SUMMARY:
Conduct a study of people who use drugs (PWUD) perceptions of and access to COVID-19 vaccines as well as reasons for vaccine hesitancy/barriers

DETAILED DESCRIPTION:
Conduct a qualitative rapid longitudinal assessment of 20 PWUD's perceptions of and access to COVID-19 vaccines as well as reasons for vaccine hesitancy/barriers. The investigators will also assess frequency and content of COVID-19 communication with peers. The investigators will also assess changes in the social network dynamics of drug use and access to illicit drugs, drug treatment, and HIV care. The brief qualitative interviews will be conducted biweekly over a period of one year. These interviews will be quickly transcribed, summarized, and provided to local and state health departments. The investigators will also use the findings from this aim to inform the proposed app and peer education pilot outlined in aims 2 & 3.

2. Development of an app provide real-time information on COVID-19 vaccine availability and nearby risk reduction resources (naloxone distribution sites, syringe exchanges, drug treatment). The app will be built for mobile download and as an online webpage. 20 PWUD will be included in this study component, split between the mobile and web-based app.

3. Develop training materials and pilot the training of 40 PWUD to promote vaccine uptake among the participants network and other community members. PWUD will be trained to become peer educators to promote COVID-19 vaccine uptake over 4 sessions. These 40 participants will be administered pre- and post-surveys as well as daily check-in questions through the app to assess effectiveness as peer educators.

ELIGIBILITY:
Inclusion Criteria:

* opioid use in prior 2 weeks

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Vaccine acceptance as assessed by the Oxford COVID-19 Vaccine Hesitancy Scale | 1 month
  Vaccine acceptance will be assessed using the Oxford COVID-19 Vaccine Hesitancy Scale, a seven-item scale that measures willingness to receive a COVID-19 vaccine. Scores ranged from 7 to 35, with higher scores indicating greater hesitancy.

CONTACTS AND LOCATIONS:
Overall Officials: Carl Latkin, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
one year after study completion
Supporting Information: Study Protocol
Time Frame: 1 year
Access Criteria: researchers